CLINICAL TRIAL: NCT04874922
Title: The Effect Birth Outcome and Diabetes Management of Planned Behavior Theory Based Education Model in Women With Gestational Diabetes
Brief Title: Gestational Diabetes Management Based on Planned Behavior Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: kocU-SDinmez
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Gestational
Keywords: Education, Nursing; Pregnancy Complications; Complications, Labor; Diabetes, Pregnancy-Induced
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications; Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: Pregnant women diagnosed with gestational diabetes will be assigned to the case and control groups in a randomized controlled manner (with simple random numbers table). Matching will be made between groups according to age and education level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): The case group will first receive standard diabetes training from the hospital. After 28-30. Diabetes training based on Planned Behavior Theory will be given three times between gestational weeks. Each training will take an average of 45 minutes. After that, the data evaluation phase will be started.
  Interventions: Behavioral: Gestational Diabetes Training Intervention based on Planned Behavior Theory
- Control Group (Other): The control group will only receive standart diabetes training from the hospital. Then, only follow-up will be done and the data will be evaluated.
  Interventions: Behavioral: Gestational Diabetes Training Intervention based on standart

INTERVENTIONS:
Behavioral: Gestational Diabetes Training Intervention based on Planned Behavior Theory — On the basis of Planned Behavior Theory, an training intervention is planned in three stages for medical nutrition, physical activity and gestational diabetes follow-up.
  Arms: Case group
Behavioral: Gestational Diabetes Training Intervention based on standart — Standard training for gestational diabetes will be given once at 28 weeks of gestation.
  Arms: Control Group

SUMMARY:
Our study was planned as a randomized controlled trial in order to determine the effect of Planned Behavior Theory based training model on diabetes management and pregnancy outcomes in women with Gestational Diabetes Mellitus.

DETAILED DESCRIPTION:
The trial will be conducted to evaluate the effectiveness of the model and to determine the impact of the Planned Behavior Theory based educational intervention on diabetes management and pregnancy outcomes.The research will be conducted in Women's Training and Research Hospitals in Istanbul. The sample group will be 70 subjects calculated by power analysis. Case and control groups will be determined by simple randomization. Sampling selection criteria; 24-28. they are pregnant women who are diagnosed with GDM between the weeks of gestation, can communicate in Turkish, are literate, have no GDM in their previous pregnancies, have a personal contact number and e-mail address, and plan to give birth at the hospital where the study will be conducted. Research data will be collected by the researcher between the 28th week of gestation and the 12th week of postpartum through the Diabetes Intention, Attitude and Behavior Questionnaire, Personal Data Collection Form, Metabolic Control Variables Form, Maternal and Infant Pregnancy Results Form. Case group; In addition to the training given in the hospital, the Training for Gestational Diabetes Based on Planned Behavior Theory will be given in three stages. Figures, percentage distributions, chi-square test, student t-test and analysis of variance will be used in the analysis of the data. As a result of the intervention made to the case group; It is expected to decrease complications due to diabetes in mothers, babies and newborns, to provide maternal metabolic control, to control the mother's weight and to shorten the duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Sample selection criteria describe pregnant women with personal contact information available who are diagnosed to have GDM between the weeks of 24-28 of their pregnancy, literate and capable of communicating in Turkish, not diagnosed to have GDM in their previous pregnancies, planning to deliver the child in the hospital where the research is to be conducted.

Exclusion Criteria:

* Not having had a cesarean delivery before.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As the study was about pregnancy, only women were included.
Enrollment: 66 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
metabolic control variables evaluation form (first) | The data of metabolic control variables of each pregnant woman at 28th gestational week will be evaluated.
  It is a form that evaluates the blood sugar, blood lipids, blood pressure, weight and insulin usage doses of pregnant women.
metabolic control variables evaluation form (second) | The data of metabolic control variables of each pregnant woman at 32nd gestational week will be evaluated.
  It is a form that evaluates the blood sugar, blood lipids, blood pressure, weight and insulin usage doses of pregnant women.
metabolic control variables evaluation form (third) | The data of metabolic control variables of each pregnant woman at her 36th gestational week will be evaluated.
  It is a form that evaluates the blood sugar, blood lipids, blood pressure, weight and insulin usage doses of pregnant women.
metabolic control variables evaluation form (fourth) | The data of metabolic control variables of each pregnant woman at her 40th gestational week will be evaluated.
  It is a form that evaluates the blood sugar, blood lipids, blood pressure, weight and insulin usage doses of pregnant women.

SECONDARY OUTCOMES:
Pregnancy Outcomes Evaluation Form for Mother and Baby | Data of each pregnant woman will be evaluated with Pregnancy Outcome Form for Mother and Baby in the postnatal period of 12 weeks.
  This form evaluates the birth information of the mother and the baby, their health conditions and birth complications.

CONTACTS AND LOCATIONS:
Overall Officials: Kafiye EROĞLU, Prof., Study Director — Koç University
Locations (1):
- Kafiye EROĞLU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blue CL, Marrero DG. Psychometric properties of the healthful eating belief scales for persons at risk of diabetes. J Nutr Educ Behav. 2006 May-Jun;38(3):134-42. doi: 10.1016/j.jneb.2006.01.010. PMID 16731447
- [Background] Blue CL, Marrero DG, Black DR. Physical activity belief scales for diabetes risk: development and psychometric testing. Health Educ Behav. 2008 Jun;35(3):316-31. doi: 10.1177/1090198106297060. Epub 2007 Jul 9. PMID 17620669
- [Background] Catalano HP, Knowlden AP, Birch DA, Leeper JD, Paschal AM, Usdan SL. Using the Theory of Planned Behavior to predict HPV vaccination intentions of college men. J Am Coll Health. 2017 Apr;65(3):197-207. doi: 10.1080/07448481.2016.1269771. Epub 2016 Dec 14. PMID 27960609
- [Background] Farmer A, Kinmonth AL, Sutton S. Measuring beliefs about taking hypoglycaemic medication among people with Type 2 diabetes. Diabet Med. 2006 Mar;23(3):265-70. doi: 10.1111/j.1464-5491.2005.01778.x. PMID 16492209
- [Background] Karacam Z, CelIk D. The prevalence and risk factors of gestational diabetes mellitus in Turkey: a systematic review and meta-analysis. J Matern Fetal Neonatal Med. 2021 Apr;34(8):1331-1341. doi: 10.1080/14767058.2019.1635109. Epub 2019 Jul 2. PMID 31220964
- [Background] Rogozinska E, Chamillard M, Hitman GA, Khan KS, Thangaratinam S. Nutritional manipulation for the primary prevention of gestational diabetes mellitus: a meta-analysis of randomised studies. PLoS One. 2015 Feb 26;10(2):e0115526. doi: 10.1371/journal.pone.0115526. eCollection 2015. PMID 25719363
- [Result] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Result] American Diabetes Association. 13. Management of Diabetes in Pregnancy: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S137-S143. doi: 10.2337/dc18-S013. PMID 29222384
- [Result] Ajzen I. The theory of planned behaviour: reactions and reflections. Psychol Health. 2011 Sep;26(9):1113-27. doi: 10.1080/08870446.2011.613995. PMID 21929476
- [Result] Akbar H, Anderson D, Gallegos D. Predicting intentions and behaviours in populations with or at-risk of diabetes: A systematic review. Prev Med Rep. 2015 Apr 14;2:270-82. doi: 10.1016/j.pmedr.2015.04.006. eCollection 2015. PMID 26844083
- [Result] Aktun HL, Uyan D, Yorgunlar B, Acet M. Gestational diabetes mellitus screening and outcomes. J Turk Ger Gynecol Assoc. 2015 Mar 1;16(1):25-9. doi: 10.5152/jtgga.2015.15081. eCollection 2015. PMID 25788845
- [Result] Ali S, Dornhorst A. Diabetes in pregnancy: health risks and management. Postgrad Med J. 2011 Jun;87(1028):417-27. doi: 10.1136/pgmj.2010.109157. Epub 2011 Mar 2. PMID 21368321
- [Result] Brown J, Alwan NA, West J, Brown S, McKinlay CJ, Farrar D, Crowther CA. Lifestyle interventions for the treatment of women with gestational diabetes. Cochrane Database Syst Rev. 2017 May 4;5(5):CD011970. doi: 10.1002/14651858.CD011970.pub2. PMID 28472859
- [Result] Coelho MCVS, Almeida CAPL, Silva ARVD, Moura LKB, Feitosa LGGC, Nunes LB. Training in diabetes education: meanings attributed by primary care nurses. Rev Bras Enferm. 2018;71(suppl 4):1611-1618. doi: 10.1590/0034-7167-2017-0792. English, Portuguese. PMID 30088631
- [Result] Griffith RJ, Alsweiler J, Moore AE, Brown S, Middleton P, Shepherd E, Crowther CA. Interventions to prevent women from developing gestational diabetes mellitus: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2020 Jun 11;6(6):CD012394. doi: 10.1002/14651858.CD012394.pub3. PMID 32526091
- [Result] Jennings CA, Vandelanotte C, Caperchione CM, Mummery WK. Effectiveness of a web-based physical activity intervention for adults with Type 2 diabetes-a randomised controlled trial. Prev Med. 2014 Mar;60:33-40. doi: 10.1016/j.ypmed.2013.12.011. Epub 2013 Dec 15. PMID 24345601
- [Result] Jones EJ, Roche CC, Appel SJ. A review of the health beliefs and lifestyle behaviors of women with previous gestational diabetes. J Obstet Gynecol Neonatal Nurs. 2009 Sep-Oct;38(5):516-26. doi: 10.1111/j.1552-6909.2009.01051.x. PMID 19883473
- [Result] Zhang C, Tobias DK, Chavarro JE, Bao W, Wang D, Ley SH, Hu FB. Adherence to healthy lifestyle and risk of gestational diabetes mellitus: prospective cohort study. BMJ. 2014 Sep 30;349:g5450. doi: 10.1136/bmj.g5450. PMID 25269649
- See also: Republic of Turkey Ministry of Health antenatal care and management guide — https://khgmsaglikhizmetleridb.saglik.gov.tr/TR,42839/dogum-oncesi-bakim-yonetim-rehberi.html
- See also: Republic of Turkey Ministry of Health-risk pregnancy care and management guide — https://khgmsaglikhizmetleridb.saglik.gov.tr/TR,42842/riskli-gebelik-yonetim-rehberi.html